CLINICAL TRIAL: NCT06371638
Title: Continuous Dexmedetomidine Infusion Reduces Postoperative Cognitive Dysfunction and Postoperative Pain in Patients Undergoing Laparatomy
Brief Title: Dexmedetomidine and Postoperative Cognitive Dysfunction (POCD)
Acronym: CODE-POCD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Udayana University (Other)
Responsible Party: Principal Investigator, Christopher Ryalino, MD, Assistant Professor, Udayana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2024-01
Record Dates: First submitted 2024-04-14; First posted 2024-04-17 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Cognitive Dysfunction; Postoperative Pain
Keywords: postoperative cognitive complications; dexmedetomidine; pain; hemodynamics
MeSH Terms: conditions — Postoperative Cognitive Complications; Pain, Postoperative; Pain | interventions — Dexmedetomidine; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patients with POCD (Experimental): MMSE was assessed 24h before surgery, 3 days after surgery, and 30 days before surgery. Subjects is considered to have POCD if the postoperative MMSE score was lower by at least 2 points compared to the preoperative score.
  Interventions: Drug: Dexmedetomidine; Drug: Sevoflurane
- Patients without POCD (Active Comparator): MMSE was assessed 24h before surgery, 3 days after surgery, and 30 days before surgery. Subjects is considered to have POCD if the postoperative MMSE score was lower by at least 2 points compared to the preoperative score.
  Interventions: Drug: Dexmedetomidine; Drug: Sevoflurane

INTERVENTIONS:
Drug: Dexmedetomidine — General anaesthesia for subjects in Group D was maintained by target-controlled infusion (TCI) dexmedetomidine (Dyck mode) with target plasma of 1 ng/ml
  Other Names: Group D
Drug: Sevoflurane — General anaesthesia for subjects in Group I was maintained by inhalation anaesthesia using sevoflurane at 0.8% concentration.
  Other Names: Group I

SUMMARY:
Postoperative cognitive dysfunction (POCD) affects all age groups and can lead to increased morbidity and more extended hospital stays. Dexmedetomidine reduces POCD by inhibiting the increase in proinflammatory cytokines IL-6 and TNF-α, and its anti-inflammatory activity contributes to its protective effect. Previous studies found that dexmedetomidine reduced POCD incidence in non-cardiac and cardiac surgery. Therefore, the goal of this study was to specifically investigate if using TCI dexmedetomidine to maintain anaesthesia in laparotomy surgeries reduces the incidence of POCD compared to inhalation anaesthesia by sevoflurane.

ELIGIBILITY:
Inclusion Criteria:

* Aged >= 18 years old
* Scheduled for laparatomy surgery

Exclusion Criteria:

* history of allergies to anaesthetic drugs
* impaired consciousness
* neurocognitive disorder
* psychiatric disorder
* mental disorder
* cerebrovascular disorders
* sick sinus syndrome
* hypoalbuminemia
* massive bleeding
* liver disease
* kidney diseases.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2024-01-07 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-07 (Actual)

PRIMARY OUTCOMES:
Postoperative cognitive dysfunction (POCD) | 48 hours postoperative
  Assessed by Mini-Mental State Examination (MMSE). Defined if there is a >= 2 points decrease compared to baseline.
Postoperative cognitive dysfunction (POCD) | 30 days postoperative
  Assessed by Mini-Mental State Examination (MMSE). Defined if there is a >= 2 points decrease compared to baseline.

SECONDARY OUTCOMES:
Intraoperative hemodynamics: mean arterial pressure (MAP) | During the course of intraoperative period.
  MAP as presented by intraoperative standard monitoring
Intraoperative hemodynamics: heart rate (HR) | During the course of intraoperative period.
  HR as presented by intraoperative standard monitoring
Postoperative pain | 1 hour postoperative
  Assessed by visual analog scale (VAS), minimum value=0 (no pain), maximum=10 (worst pain)
Postoperative pain | 12 hours postoperative
  Assessed by visual analog scale (VAS), minimum value=0 (no pain), maximum=10 (worst pain)
Postoperative pain | 24 hours postoperative
  Assessed by visual analog scale (VAS), minimum value=0 (no pain), maximum=10 (worst pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Prof. Ngoerah General Hospital, Denpasar, Bali, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
Data is available for other researchers upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Start: once study is published Until: 1-year after publication